CLINICAL TRIAL: NCT02659943
Title: T Cells Expressing a Fully-Human Anti-CD19 Chimeric Antigen Receptor for Treating B-cell Malignancies
Brief Title: T Cells Expressing a Fully-human AntiCD19 Chimeric Antigen Receptor for Treating B-cell Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, James Kochenderfer, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 160054; 16-C-0054
Record Dates: First submitted 2016-01-20; First posted 2016-01-21 (Estimated); Results first posted 2021-05-04 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-03

CONDITIONS: Lymphoma, B-Cell; Lymphoma, Non-hodgkins
Keywords: Gene Therapy; Adoptive T Cell Therapy; Allogeneic Stem Cell Transplantation; T-cell infusion; Residual Malignancy
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Non-Hodgkin | interventions — Automobiles; Cyclophosphamide; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- LEVEL 1 - Participants Who Received 0.66x10^6 CAR T Cells Only (Experimental): LEVEL 1 - participants who received - 0.66x10^6 Chimeric Antigen Receptor (CAR) T cells only
  Interventions: Biological: Anti-cluster of differentiation 19 (CD19)-Chimeric Antigen Receptor (CAR) T cells
- LEVEL 1 Foll/by LEVEL 2-Participants Who Received - 0.66x10^6 CAR T Cells Foll/by 2x10^6 CAR T Cells (Experimental): LEVEL 1 followed by LEVEL 2 - participants who received - 0.66x10^6 Chimeric Antigen Receptor (CAR) T cells followed by 2x10^6 CAR T cells
  Interventions: Biological: Anti-cluster of differentiation 19 (CD19)-Chimeric Antigen Receptor (CAR) T cells; Drug: Cyclophosphamide; Drug: Fludarabine
- LEVEL 1 Foll/by LEVEL 3 - Participants Who Received 0.66x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells (Experimental): LEVEL 1 followed by LEVEL 3 - participant who received - 0.66x10^6 Chimeric Antigen Receptor (CAR) T cells followed by 6x10^6 CAR T cells
  Interventions: Biological: Anti-cluster of differentiation 19 (CD19)-Chimeric Antigen Receptor (CAR) T cells; Drug: Cyclophosphamide; Drug: Fludarabine
- LEVEL 2 - Participants Who Received 2x10^6 CAR T Cells Only (Experimental): LEVEL 2 - participants who received - 2x10^6 Chimeric Antigen Receptor (CAR) T cells only
  Interventions: Biological: Anti-cluster of differentiation 19 (CD19)-Chimeric Antigen Receptor (CAR) T cells
- LEVEL 2 Followed by LEVEL 3-Participants Who Received 2x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells (Experimental): LEVEL 2 followed by LEVEL 3 - participants who received - 2x10^6 Chimeric Antigen Receptor (CAR) T cells followed by 6x10^6 CAR T cells
  Interventions: Biological: Anti-cluster of differentiation 19 (CD19)-Chimeric Antigen Receptor (CAR) T cells; Drug: Cyclophosphamide; Drug: Fludarabine
- LEVEL 3 - Participants Who Received 6x10^6 CAR T Cells Only (Experimental): LEVEL 3 - participants who received - 6x10^6 Chimeric Antigen Receptor (CAR) T cells only
  Interventions: Biological: Anti-cluster of differentiation 19 (CD19)-Chimeric Antigen Receptor (CAR) T cells

INTERVENTIONS:
Biological: Anti-cluster of differentiation 19 (CD19)-Chimeric Antigen Receptor (CAR) T cells — Dose-escalation trial starting dose: 0.66x10^6 CAR+ T cells/kg(weight based dosing)(up to a maximum dose of 18x10^6 CAR+ T cells/kg) infuse on day 0
Drug: Cyclophosphamide — 300 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3
  Other Names: Cytoxan
  Arms: LEVEL 1 Foll/by LEVEL 2-Participants Who Received - 0.66x10^6 CAR T Cells Foll/by 2x10^6 CAR T Cells; LEVEL 1 Foll/by LEVEL 3 - Participants Who Received 0.66x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells; LEVEL 2 Followed by LEVEL 3-Participants Who Received 2x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells
Drug: Fludarabine — 30 mg/m^2 intravenous (IV) infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4,and -3
  Other Names: Fludara
  Arms: LEVEL 1 Foll/by LEVEL 2-Participants Who Received - 0.66x10^6 CAR T Cells Foll/by 2x10^6 CAR T Cells; LEVEL 1 Foll/by LEVEL 3 - Participants Who Received 0.66x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells; LEVEL 2 Followed by LEVEL 3-Participants Who Received 2x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells

SUMMARY:
Background:

The immune system fights infection and can affect cancer cells. T cells are white blood cells that are a major part of the immune system. T cells can destroy tumors. Researchers want to try to manipulate the immune system to better recognize and kill tumor cells.

Objective:

To test the safety of giving T cells expressing a novel fully-human anti-cluster of differentiation 19 (CD19) chimeric antigen receptor (CAR) to people with advanced B-cell cancer.

Eligibility:

People ages 18-73 with a B-cell cancer that has not been controlled by other therapies.

Design:

Participants will be screened with:

Physical exam

Blood and urine tests

Heart tests

Bone marrow sample taken

Scans in machines that take pictures

Participants will have apheresis. Blood is removed through a needle in an arm. T cells are removed. The rest of the blood is returned through a needle in the other arm.

The cells will be changed in a laboratory.

Participants will get 2 chemotherapy drugs over 3 days.

Two days later, participants will check into the hospital. They will get an intravenous (IV) catheter in an arm or chest vein. They will get the T cells through the IV in 1 infusion.

After this, participants will stay in the hospital for at least 9 days and stay nearby for 2 weeks. Then they will have blood tests and see a doctor.

Participants will have visits 6 visits for 1 year after the infusion. Some may have more follow-up visits.

Participants may samples taken of spinal fluid, bone marrow, and tumors.

...

DETAILED DESCRIPTION:
Background:

* Improved treatments for a variety of treatment-resistant B-cell malignancies including Bcell lymphomas and chronic lymphocytic leukemia (CLL), are needed.
* A particular need is development of new treatments for chemotherapy-refractory B-cell malignancies.
* T cells can be genetically modified to express chimeric antigen receptors (CARs) that specifically target malignancy-associated antigens.
* Autologous T cells genetically modified to express CARs targeting the B-cell antigen cluster of differentiation 19 (CD19) have caused complete remissions in a small number of patients with leukemia or lymphoma. These results demonstrate that anti-CD19 CAR-expressing T cells have antimalignancy activity in humans.
* The vast majority of B-cell malignancies express CD19.
* CD19 is not expressed by normal cells except for B cells.
* We have constructed a novel fully-human anti-CD19 CAR that can specifically recognize CD19-expressing target cells in vitro and eradicate CD19-expressing tumors in mice.
* This fully-human CAR targeting CD19 has not been tested in humans before.
* Possible toxicities include cytokine-associated toxicities such as fever, hypotension, and neurological toxicities. Elimination of normal B cells is probable, and unknown toxicities are also possible.

Objectives:

Primary

-Determine the safety and feasibility of administering T cells expressing a novel fully-human anti-CD19 CAR to patients with advanced B-cell malignancies.

Secondary

* Evaluate the in vivo persistence and peak blood levels of anti-CD19 CAR T cells after initial and repeated CAR T-cell infusions. CAR T-cell blood levels will be compared retrospectively to results with an anti-CD19 CAR containing an antigen-recognition moiety derived from a murine antibody.
* Assess for evidence of anti-malignancy activity by anti-CD19 CAR T cells
* Assess the impact of repeated CAR T-cell infusions on residual malignancy after an initial CAR T-cell infusion.
* Assess the immunogenicity of the CAR used in this protocol.

Eligibility:

* Patients must have any B-cell lymphoma, or CLL/small lymphocytic lymphoma (SLL). Lower grade lymphomas transformed to DLBCL are potentially eligible as is primary mediastinal B-cell lymphoma and all other subtypes of Diffuse large B-cell lymphoma (DLBCL).
* Patients must have malignancy that is measurable on a computed tomography (CT) scan or by flow cytometry of bone marrow or blood.
* Patients must have a creatinine of 1.4 mg/dL or less and a normal cardiac ejection fraction.
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 is required.
* No active infections are allowed including any history of hepatitis B or hepatitis C.
* Absolute neutrophil count greater than or equal to1000/microliter, platelet count greater than or equal to 45,000/microliter, hemoglobin greater than or equal to 8g/dL
* Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less or equal to 3 times the upper limit of the institutional normal unless liver involvement by malignancy is demonstrated.
* At least 14 days must elapse between the time of any prior systemic treatment (including corticosteroids) and initiation of protocol enrollment.
* The patients malignancy will need to be assessed for CD19 expression by flow cytometry or immunohistochemistry performed at the National Institutes of Health (NIH). If unstained, paraffinembedded bone marrow or lymphoma sections are available from prior biopsies, these can be used to determine CD19 expression by immunohistochemistry; otherwise, patients will need to come to the NIH for a biopsy to determine CD19 expression. The sample for CD19 expression can come from a biopsy obtained at any time before enrollment.
* Patients who have never had an allogeneic hematopoietic stem cell transplant are potentially eligible.

Design:

* This is a phase I dose-escalation trial
* Patients will undergo leukapheresis
* T-cells obtained by leukapheresis will be genetically modified to express an anti-CD19 CAR
* Patients will receive a lymphocyte-depleting chemotherapy conditioning regimen with the intent of enhancing the activity of the infused anti-CD19-CAR-expressing T cells.
* The chemotherapy conditioning regimen is cyclophosphamide 300 mg/m(2) daily for 3 days and fludarabine 30 mg/m(2) daily for 3 days. Fludarabine will be given on the same days as the cyclophosphamide.
* Two days after the chemotherapy ends, patients will receive an infusion of anti-CD19-CAR-expressing T cells.
* The initial dose level of this dose-escalation trial will be 0.66x10(6) CAR+ T cells/kg of recipient bodyweight.
* The cell dose administered will be escalated until a maximum tolerated dose is determined.
* Following the T-cell infusion, there is a mandatory 9-day inpatient hospitalization to monitor for toxicity.
* Outpatient follow-up is planned for 2 weeks, and 1, 2, 3, 6, 9, and 12 months after the CAR T-cell infusion. Long-term gene-therapy follow-up consisting of yearly visits to a doctor near the patient s home for 4 more years and then yearly telephone contact for 10 additional years will be required.
* Repeat treatments consisting of the conditioning chemotherapy followed by a CAR T-cell infusion are planned for eligible patients with any best responses except continuing complete remission or progressive malignancy.
* Re-enrollment will be allowed for a small number of subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Malignancy criteria:

  * Patients with the following malignancies are potentially eligible: any B-cell lymphoma, and chronic lymphocytic leukemia (CLL). Patients with indolent malignancies that have transformed to diffuse large B-cell lymphoma are eligible.
  * Clear cluster of differentiation 19 (CD19) expression must be uniformly detected on 75% or more of malignant cells from either bone marrow or a leukemia or lymphoma mass by flow cytometry or immunohistochemistry. These assays must be performed at the National Institutes of Health. It is preferable but not required that the specimen used for CD19 determination comes from a sample that was obtained after the patient's most recent treatment. If paraffin embedded unstained samples of bone marrow involved with malignancy or a lymphoma mass are available, these can be shipped to the National Institutes of Health (NIH) for CD19 staining; otherwise, new biopsies will need to be performed for determination of CD19 expression.
  * Diffuse large B-cell lymphoma (DLBCL) patients must have received at least two prior chemotherapy-containing regimens at least one of which must have contained doxorubicin and a monoclonal antibody. Follicular lymphoma patients must have received at least 2 prior regimens including at least 1 regimen with chemotherapy. All other lymphoma and leukemia patients must have had at least 1 prior chemotherapy-containing regimen. All patients with CLL or small lymphocytic lymphoma must have had prior treatment with ibrutinib or another signal transduction inhibitor.
  * Patients must have measurable malignancy as defined by at least one of the criteria below.

    * Lymphoma or leukemia masses that are measurable (minimum 1.5 cm in largest diameter) by computed tomography (CT) scan is required for all diagnoses except CLL. All masses must be less than 10 cm in the largest diameter.
    * For a lymphoma mass to count as measurable malignancy, it must have abnormally increased metabolic activity when assessed by positron emission tomography (PET) scan.
    * For CLL and lymphoma with only bone marrow involvement no mass is necessary, but if a mass is not present, bone marrow malignancy must be detectable by flow cytometry in lymphoma and CLL.
* Other inclusion criteria:

  * Greater than or equal to 18 years of age and less than or equal to age 73.
  * Able to understand and sign the Informed Consent Document.
  * Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0-1
  * Room air oxygen saturation of 92% or greater
  * Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for four months after receiving the preparative regimen.
  * Women of child bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the preparative chemotherapy on the fetus. Women of child-bearing potential are defined as all women except women who are post-menopausal or who have had a hysterectomy. Postmenopausal will be defined as women over the age of 55 who have not had a menstrual period in at least 1 year.
  * Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune -competence and thus are less responsive to the experimental treatment and more susceptible to its toxicities.)
  * Patients with a known history of hepatitis B or hepatitis C are not eligible due to the risk of re-activation of hepatitis after prolonged B-cell depletion due to anti-CD19 CAR T cells.
  * Seronegative for hepatitis B antigen, positive hepatitis B tests can be further evaluated by confirmatory tests, and if confirmatory tests are negative, the patient can be enrolled. Patients with a known history of hepatitis B are not eligible.
  * Seronegative for hepatitis C antibody unless antigen negative. If hepatitis C antibody test is positive, then patients must be tested for the presence of ribonucleic acid (RNA) by reverse transcription polymerase chain reaction (RT-PCR) and be hepatitis C virus (HCV) RNA negative. Patients with a known history of hepatitis C are not eligible.
  * Absolute neutrophil count greater than or equal to 1000/mm(3) without the support of filgrastim or other growth factors.
  * Platelet count greater than or equal to 45,000/mm(3) without transfusion support
  * Hemoglobin greater than 8.0 g/dl.
  * Less than 5% malignant cells in the peripheral blood leukocytes
  * Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less or equal to 3 times the upper limit of the institutional normal unless liver involvement by malignancy is demonstrated.
  * Serum creatinine less than or equal to 1.4 mg/dL.
  * Total bilirubin less than or equal to 2.0 mg/dl.
  * At least 14 days must have elapsed since any prior systemic therapy prior to apheresis and prior to the initiation of chemotherapy (including systemic corticosteroids at any dose). Because this protocol requires collection of autologous blood cells by leukapheresis in order to prepare CAR T cells, systemic anti-malignancy therapy including systemic corticosteroid therapy of any dose are not allowed within 14 days prior to the required leukapheresis. NOTE: Because of the long half-life and potential to affect CAR T cells, 60 days must elapse from the time of administration of anti-Programmed cell death protein 1 (PD-1) or anti-Programmed death-ligand 1 (PD-L1) antibodies or other agents that in the opinion of the PI can stimulate immune activity and infusion of CAR T cells.
  * Normal cardiac ejection fraction (greater than or equal to 55% by echocardiography) and no evidence of hemodynamically significant pericardial effusion as determined by an echocardiogram within 4 weeks of the start of the treatment protocol.
  * Patients must not take corticosteroids including prednisone, dexamethasone or any other corticosteroid for 14 days before apheresis and CAR T-cell infusion. Patients must also not take corticosteroids at doses higher than 5 mg/day of prednisone or equivalent at any time after the CAR T cell infusion.
  * Patients who have been treated on other protocols of genetically-modified T cells at the NIH only are potentially eligible under these conditions:

    * At least 6 months have elapsed since the last genetically-modified T-cell therapy that the patient received and there is no evidence of replication-competent retroviruses (evidence must be provided from prior NIH gene-therapy protocol Principal Investigator) and persisting genetically-modified T cells are not detectable in the patient's blood (evidence must be provided by prior NIH gene-therapy protocol Principal Investigator).

EXCLUSION CRITERIA:

* Patients that require urgent therapy due to tumor mass effects or spinal cord compression.
* Patients that have active hemolytic anemia.
* Patients with second malignancies in addition to their B-cell malignancy are not eligible if the second malignancy has required treatment (including maintenance therapy) within the past 4 years or is not in complete remission. There are two exceptions to this criterion: successfully treated non-metastatic basal cell or squamous cell skin carcinoma.
* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
* Active uncontrolled systemic infections (defined as infections causing fevers and infections requiring intravenous antibiotics when intravenous antibiotics have been administered for less than 72 hours), active coagulation disorders or other major uncontrolled medical illnesses of the cardiovascular, respiratory, endocrine, renal, gastrointestinal, genitourinary or immune system, history of myocardial infarction, history of ventricular tachycardia or ventricular fibrillation, active cardiac arrhythmias (active atrial fibrillation is not allowed, resolved atrial fibrillation not requiring current treatment is allowed (anticoagulants count as current treatment) ), active obstructive or restrictive pulmonary disease, active autoimmune diseases such as rheumatoid arthritis.
* Patients will not be seen for screening appointments or enrolled on the protocol if they have been hospitalized within the 7 days prior to the screening appointment or the date of protocol enrollment.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* Systemic corticosteroid steroid therapy of any dose is not allowed within 14 days prior to the required leukapheresis, or the initiation of the conditioning chemotherapy regimen. Corticosteroid creams, ointments, and eye drops are allowed.
* History of severe immediate hypersensitivity reaction to any of the agents used in this study.
* Patients with current central nervous system (CNS) involvement by malignancy (either by imaging or cerebrospinal fluid involvement or biopsy-proven).

Ages: 18 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-01-21 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James N Kochenderfer, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-C-0054.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Enrolled But Not Treated: Participants who were enrolled but not treated.
Period: Overall Study
Arm/Group | LEVEL 1 - Participants Who Received 0.66x10^6 CAR T Cells Only | LEVEL 1 Foll/by LEVEL 2-Participants Who Received - 0.66x10^6 CAR T Cells Foll/by 2x10^6 CAR T Cells | LEVEL 1 Foll/by LEVEL 3 - Participants Who Received 0.66x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells | LEVEL 2 - Participants Who Received 2x10^6 CAR T Cells Only | LEVEL 2 Followed by LEVEL 3-Participants Who Received 2x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells | LEVEL 3 - Participants Who Received 6x10^6 CAR T Cells Only | Participants Enrolled But Not Treated
Started | 3 | 2 | 1 | 4 | 2 | 9 | 6
Completed | 2 | 0 | 0 | 1 | 0 | 4 | 0
Not Completed | 1 | 2 | 1 | 3 | 2 | 5 | 6
Not completed — Switched to alternative treatment | 1 | 1 | 0 | 2 | 1 | 0 | 1
Not completed — Disease progression on study | 0 | 1 | 1 | 1 | 1 | 4 | 0
Not completed — Patient's condition per principal investigator | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Ineligible | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — No longer meets eligibility | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — No treatment, per protocol | 0 | 0 | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Baseline data was collected and reported here for the participants enrolled but not treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | LEVEL 1 - Participants Who Received 0.66x10^6 CAR T Cells Only | LEVEL 1 Foll/by LEVEL 2-Participants Who Received - 0.66x10^6 CAR T Cells Foll/by 2x10^6 CAR T Cells | LEVEL 1 Foll/by LEVEL 3 - Participants Who Received 0.66x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells | LEVEL 2 - Participants Who Received 2x10^6 CAR T Cells Only | LEVEL 2 Followed by LEVEL 3-Participants Who Received 2x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells | LEVEL 3 - Participants Who Received 6x10^6 CAR T Cells Only | Participants Enrolled But Not Treated | Total
Number analyzed (Participants) | 3 | 2 | 1 | 4 | 2 | 9 | 6 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 0 | 3 | 1 | 6 | 4 | 18
  >=65 years | 1 | 0 | 1 | 1 | 1 | 3 | 2 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (10.14) | 50.35 (3.04) | 68.6 (0) | 57.2 (8.61) | 65 (5.09) | 57.11 (10.8) | 52.98 (16.32) | 56.55 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 0 | 0 | 5 | 2 | 11
  Male | 1 | 1 | 0 | 4 | 2 | 4 | 4 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 2 | 1 | 4 | 2 | 7 | 6 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 1 | 1 | 4 | 2 | 8 | 6 | 25
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 1 | 4 | 2 | 9 | 6 | 27
Prior Lines of Therapy [Count of Participants; unit: Participants]
  1 Line of therapy | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  2 Lines of therapy | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 6
  3 Lines of therapy | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 4
  4 Lines of therapy | 1 | 0 | 1 | 1 | 0 | 4 | 0 | 7
  5 Lines of therapy | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3
  6 Lines of therapy | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 3
  9 Lines of therapy | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Lymphoma Type [Count of Participants; unit: Participants]
  DLBCL | 1 | 0 | 0 | 1 | 1 | 4 | 3 | 10
  DLBCL transformed from follicular lymphoma | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
  DLBCL, double-hit | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 3
  DLBCL, triple-hit | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Mantle-cell lymphoma | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3
  Follicular lymphoma | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 3
  Burkitt lymphoma | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  CLL/DLBCL | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  ALL | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Enrolled Participants Who Actually Get Treated
Description: Percentage of participants enrolled who received treatment with Chimeric Antigen Receptor (CAR) T cells, Fludarabine and cyclophosphamide.
Time Frame: 4-5 weeks after the first dose
Population: Data is combined for this outcome measure because it is not possible to draw firm conclusions from the small number of participants in each dose level; the data drawn from the overall participant population through the course of the trial is much more meaningful and conclusive. 26/27 participants were analyzed because one participant was enrolled and cells were collected, then came off study because of ineligibility and re-enrolled much later and did receive cells at that time.
Measure: Number; unit: percentage of participants
Groups:
- All Participants: All participants who received Biological/Vaccine: Anti-cluster of differentiation 19 (CD19)-Chimeric Antigen Receptor (CAR) T cells Dose-escalation trial starting dose: 0.66x10^6 CAR+ T cells/kg (weight-based dosing) (up to a maximum dose of 18x10^6 CAR+ T cells/kg) infuse on day 0 Drug: Cyclophosphamide 300 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 Drug: Fludarabine 30 mg/m^2 intravenous (IV) infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3
Arm/Group | All Participants
Number analyzed (Participants) | 26
percentage of participants | 76.9

2. Secondary Outcome: Number of Participants Who Had a Best Response of Complete Remission (CR), Partial Remission (PR), Stable Disease (SD), and Progressive Disease (PD)
Description: Response was assessed by the Revised Response Criteria for Malignant Lymphoma, and Recommendations for Initial Evaluation, Staging, and Response Assessment of Hodgkin and Non-Hodgkin Lymphoma: The Lugano Classification. Complete Remission is complete disappearance of all detectable clinical evidence of disease. Partial Remission is ≥50% decrease in sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses. Progressive Disease is ≥50% increase from nadir in the sum of the products of at least two lymph nodes, or if a single node is involved at least a 50% increase in the product of the diameters of this one node. Stable Disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease.
Time Frame: 30 days post Chimeric Antigen Receptor (CAR) T-cells up to 5 years
Population: 6 participants were enrolled but not treated and one participant was enrolled and cells were collected, then came off study because of ineligibility and re-enrolled much later and did receive cells at that time.
Measure: Count of Participants; unit: Participants
Arm/Group | LEVEL 1 - Participants Who Received 0.66x10^6 CAR T Cells Only | LEVEL 1 Foll/by LEVEL 2-Participants Who Received - 0.66x10^6 CAR T Cells Foll/by 2x10^6 CAR T Cells | LEVEL 1 Foll/by LEVEL 3 - Participants Who Received 0.66x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells | LEVEL 2 - Participants Who Received 2x10^6 CAR T Cells Only | LEVEL 2 Followed by LEVEL 3-Participants Who Received 2x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells | LEVEL 3 - Participants Who Received 6x10^6 CAR T Cells Only
Number analyzed (Participants) | 3 | 2 | 1 | 4 | 2 | 9
Participants
  Complete Remission After First Re-Treatment | 0 | 0 | 1 | 0 | 0 | 0
  Complete Remission After Second Re-Treatment | 0 | 0 | 0 | 0 | 0 | 0
  Partial Remission After Second Re-Treatment | 0 | 1 | 0 | 0 | 1 | 0
  Stable Disease After First Re-Treatment | 0 | 0 | 0 | 0 | 1 | 0
  Stable Disease After Second Re-Treatment | 0 | 0 | 0 | 0 | 1 | 0
  Stable Disease After Third Re-Treatment | 0 | 0 | 0 | 0 | 1 | 0
  Progressive Disease After Second Re-Treatment | 0 | 1 | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With a Duration of Best Response in Months
Description: Best Response defined as the first documentation of response was assessed by the Revised Response Criteria for Malignant Lymphoma, and Recommendations for Initial Evaluation, Staging, and Response Assessment of Hodgkin and Non-Hodgkin Lymphoma: The Lugano Classification.
Time Frame: Response duration is the time from first documentation of response, which is one month after cell infusion in all participants, until progression, initiation of off-study treatment or the last documentation on ongoing response, approx. one month -5 years.
Population: No participants were analyzed in the participants enrolled but not treated Arm/Group, thus the table is not included.
Measure: Count of Participants; unit: Participants
Arm/Group | LEVEL 1 - Participants Who Received 0.66x10^6 CAR T Cells Only | LEVEL 1 Foll/by LEVEL 2-Participants Who Received - 0.66x10^6 CAR T Cells Foll/by 2x10^6 CAR T Cells | LEVEL 1 Foll/by LEVEL 3 - Participants Who Received 0.66x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells | LEVEL 2 - Participants Who Received 2x10^6 CAR T Cells Only | LEVEL 2 Followed by LEVEL 3-Participants Who Received 2x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells | LEVEL 3 - Participants Who Received 6x10^6 CAR T Cells Only
Number analyzed (Participants) | 3 | 2 | 1 | 4 | 2 | 9
Participants
  Stable Disease - 1 Month | 0 | 0 | 0 | 2 | 0 | 1
  Stable Disease - 1 Month (first of two treatments) | 0 | 1 | 0 | 0 | 0 | 0
  Stable Disease - 1 Month After First Re-Treatment | 0 | 0 | 0 | 0 | 1 | 0
  Stable Disease - 2 Months (first of three treatments) | 0 | 0 | 0 | 0 | 1 | 0
  Stable Disease - 2 Months After Second Re-Treatment | 0 | 0 | 0 | 0 | 1 | 0
  Partial Remission - 1 Month After First Re-Treatment | 0 | 1 | 0 | 0 | 1 | 0
  Partial Remission - 2 months | 0 | 0 | 0 | 0 | 0 | 2
  Partial Remission - 3 Months | 1 | 0 | 0 | 0 | 0 | 0
  Complete Remission - 4 Months (first of two treatments) | 0 | 1 | 0 | 0 | 0 | 0
  Progressive Disease - After first Re-treatment | 0 | 1 | 0 | 0 | 0 | 0
  Complete Remission - 40 Months (first of two treatments) | 0 | 0 | 1 | 0 | 0 | 0
  Complete Remission - 5 Months After First Re-Treatment | 0 | 0 | 1 | 0 | 0 | 0
  Complete Remission - 6 Months | 0 | 0 | 0 | 1 | 0 | 0
  Complete Remission - 6 Months (first of two treatments) | 0 | 0 | 0 | 0 | 1 | 0
  Complete Remission - 29+ Months | 0 | 0 | 0 | 0 | 0 | 1
  Complete Remission - 35+ Months | 0 | 0 | 0 | 1 | 0 | 3
  Complete Remission - 45+ Months | 2 | 0 | 0 | 0 | 0 | 0
  Progressive Disease | 0 | 0 | 0 | 0 | 0 | 1

4. Secondary Outcome: Number of Participants That Had Any Grade 2, 3, 4 and 5 Adverse Events
Description: Adverse Events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). Grade1 is mild, Grade 2 is moderate, Grade 3 is severe, Grade 4 is life-threatening or disabling, and Grade 5 is fatal.
Time Frame: Date treatment consent signed to date off study, approximately 49 months and 19 days.
Population: as for outcome 2
Measure: Number; unit: Adverse events
Arm/Group | LEVEL 1 - Participants Who Received 0.66x10^6 CAR T Cells Only | LEVEL 1 Foll/by LEVEL 2-Participants Who Received - 0.66x10^6 CAR T Cells Foll/by 2x10^6 CAR T Cells | LEVEL 1 Foll/by LEVEL 3 - Participants Who Received 0.66x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells | LEVEL 2 - Participants Who Received 2x10^6 CAR T Cells Only | LEVEL 2 Followed by LEVEL 3-Participants Who Received 2x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells | LEVEL 3 - Participants Who Received 6x10^6 CAR T Cells Only
Number analyzed (Participants) | 3 | 2 | 1 | 4 | 2 | 9
Adverse events
  < Grade 2 | 2 | 2 | 1 | 3 | 2 | 6
  Grade 2 | 0 | 0 | 0 | 1 | 0 | 2
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Median Peak Chimeric Antigen Receptor (CAR) T Cells Level for Participants Treated
Description: A quantitative polymerase chain reaction (PCR) assay or a flow cytometry assay will be used to quantitate Chimeric Antigen Receptor (CAR) + T cells. The absolute number of CAR+ peripheral blood mononuclear cells (PBMC) will be estimated by multiplying the percentage of CAR+ PBMC determined by PCR by the absolute number of lymphocytes plus monocytes per microliter of blood.
Time Frame: All post-infusion time-points up to at least 2 months after infusion, and CAR+ T cell analysis will continue until the CAR+ T cell level drops to undetectable levels unless a stable low level of CAR+ T cells is present at more than 3 years after infusion.
Population: as for outcome 2
Measure: Median (Full Range); unit: CAR+cell/microliter of blood
Arm/Group | LEVEL 1 - Participants Who Received 0.66x10^6 CAR T Cells Only | LEVEL 1 Foll/by LEVEL 2-Participants Who Received - 0.66x10^6 CAR T Cells Foll/by 2x10^6 CAR T Cells | LEVEL 1 Foll/by LEVEL 3 - Participants Who Received 0.66x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells | LEVEL 2 - Participants Who Received 2x10^6 CAR T Cells Only | LEVEL 2 Followed by LEVEL 3-Participants Who Received 2x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells | LEVEL 3 - Participants Who Received 6x10^6 CAR T Cells Only
Number analyzed (Participants) | 3 | 2 | 1 | 4 | 2 | 9
CAR+cell/microliter of blood | 42 [31 to 606] | 6 [1 to 33] | 4 [NA to NA] — Not available for second cell infusion. | 36 [11 to 1258] | 6 [0 to 25] | 87 [28 to 2216]

6. Secondary Outcome: Number of Participants Who Had a Second or Third Infusion of Chimeric Antigen Receptor (CAR)+ T Cells
Description: Number of participants who had a second or third Infusion Chimeric Antigen Receptor (CAR)+ T cells. Participants were eligible for a subsequent CAR T-cell infusion if the response at one month after CAR T-cell infusion was partial remission (PR) or stable disease (SD). Participants could also receive a subsequent CAR T-cell infusion if the response was complete remission (CR) but the malignancy later relapsed. CR, PR, and SD was assessed by the Revised Response Criteria for Malignant Lymphoma, and Recommendations for Initial Evaluation, Staging, and Response Assessment of Hodgkin and Non-Hodgkin Lymphoma: The Lugano Classification. Complete Remission is complete disappearance of all detectable clinical evidence of disease. Partial Remission is ≥50% decrease in sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses. Stable Disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease.
Time Frame: Participants could receive subsequent cell infusions any time 1 month after CAR T-cell infusion until 5 years after cell infusion.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | LEVEL 1 - Participants Who Received 0.66x10^6 CAR T Cells Only | LEVEL 1 Foll/by LEVEL 2-Participants Who Received - 0.66x10^6 CAR T Cells Foll/by 2x10^6 CAR T Cells | LEVEL 1 Foll/by LEVEL 3 - Participants Who Received 0.66x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells | LEVEL 2 - Participants Who Received 2x10^6 CAR T Cells Only | LEVEL 2 Followed by LEVEL 3-Participants Who Received 2x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells | LEVEL 3 - Participants Who Received 6x10^6 CAR T Cells Only
Number analyzed (Participants) | 3 | 2 | 1 | 4 | 2 | 9
Participants
  Second infusion | 0 | 2 | 1 | 0 | 1 | 0
  Third infusion | 0 | 0 | 0 | 0 | 1 | 0

7. Secondary Outcome: Number of Participants Who Had Anti-Lymphoma Activity
Description: Depending on the type of disease, we use PET/CT imaging, tumor biopsies as well as bone marrow biopsies using immunohistochemistry and flow cytometry.
Time Frame: 14 days up to 5 years post cell infusion.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | LEVEL 1 - Participants Who Received 0.66x10^6 CAR T Cells Only | LEVEL 1 Foll/by LEVEL 2-Participants Who Received - 0.66x10^6 CAR T Cells Foll/by 2x10^6 CAR T Cells | LEVEL 1 Foll/by LEVEL 3 - Participants Who Received 0.66x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells | LEVEL 2 - Participants Who Received 2x10^6 CAR T Cells Only | LEVEL 2 Followed by LEVEL 3-Participants Who Received 2x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells | LEVEL 3 - Participants Who Received 6x10^6 CAR T Cells Only
Number analyzed (Participants) | 3 | 2 | 1 | 4 | 2 | 9
Participants | 3 | 2 | 1 | 2 | 1 | 6

8. Secondary Outcome: Number of Participants With Evidence of Immunogenicity of the Chimeric Antigen Receptor (CAR) T-cell Product
Description: Enzyme-linked spot (ELISPOT) assays were performed to look for anti-CAR T-cell responses.
Time Frame: 9 days to 6 weeks after CAR T-cell infusion
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | LEVEL 1 - Participants Who Received 0.66x10^6 CAR T Cells Only | LEVEL 1 Foll/by LEVEL 2-Participants Who Received - 0.66x10^6 CAR T Cells Foll/by 2x10^6 CAR T Cells | LEVEL 1 Foll/by LEVEL 3 - Participants Who Received 0.66x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells | LEVEL 2 - Participants Who Received 2x10^6 CAR T Cells Only | LEVEL 2 Followed by LEVEL 3-Participants Who Received 2x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells | LEVEL 3 - Participants Who Received 6x10^6 CAR T Cells Only
Number analyzed (Participants) | 3 | 2 | 1 | 4 | 2 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0

9. Other Pre Specified Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 49 months and 19 days.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | LEVEL 1 - Participants Who Received 0.66x10^6 CAR T Cells Only | LEVEL 1 Foll/by LEVEL 2-Participants Who Received - 0.66x10^6 CAR T Cells Foll/by 2x10^6 CAR T Cells | LEVEL 1 Foll/by LEVEL 3 - Participants Who Received 0.66x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells | LEVEL 2 - Participants Who Received 2x10^6 CAR T Cells Only | LEVEL 2 Followed by LEVEL 3-Participants Who Received 2x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells | LEVEL 3 - Participants Who Received 6x10^6 CAR T Cells Only
Number analyzed (Participants) | 3 | 2 | 1 | 4 | 2 | 9
Participants | 3 | 2 | 1 | 4 | 2 | 9

10. Other Pre Specified Outcome: MTD
Description: The maximum tolerated dose is the dose at which a maximum of 1 of 6 patients has a dose limiting toxicity (DLT- Grade 3 toxicities possibly or probably related to toxicities possibly or probably related to either the anti-CD19 CAR T cells or the fludarabine and cyclophosphamide chemotherapy and lasting more than 7 days . Grade 4 toxicities possibly or probably related to the study interventions.).
Time Frame: Within 60 days of Chimeric Antigen Receptor (CAR) T cells infusion
Measure: Number; unit: T-cells/kg
Arm/Group | All Participants
Number analyzed (Participants) | 20
T-cells/kg | NA — The maximum tolerated dose for this protocol was not reached. 6 participants were enrolled but not treated and one participant was enrolled and cells were collected, then came off study because of ineligibility and re-enrolled much later and did receive cells at that time.

11. Other Pre Specified Outcome: Number of Participants With a Dose-Limiting Toxicity (DLT)
Description: Number of participants with DLT's defined as follows: Grade 3 toxicities possibly or probably related to toxicities possibly or probably related to either the anti-CD19 CAR T cells or the fludarabine and cyclophosphamide chemotherapy and lasting more than 7 days. Grade 4 toxicities possibly or probably related to the study interventions.
Time Frame: Within 60 days of Chimeric Antigen Receptor (CAR) T cells infusion
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | LEVEL 1 - Participants Who Received 0.66x10^6 CAR T Cells Only | LEVEL 1 Foll/by LEVEL 2-Participants Who Received - 0.66x10^6 CAR T Cells Foll/by 2x10^6 CAR T Cells | LEVEL 1 Foll/by LEVEL 3 - Participants Who Received 0.66x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells | LEVEL 2 - Participants Who Received 2x10^6 CAR T Cells Only | LEVEL 2 Followed by LEVEL 3-Participants Who Received 2x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells | LEVEL 3 - Participants Who Received 6x10^6 CAR T Cells Only
Number analyzed (Participants) | 3 | 2 | 1 | 4 | 2 | 9
Participants | 1 | 0 | 0 | 2 | 0 | 1

12. Other Pre Specified Outcome: Maximum Feasible Dose
Description: Maximum feasible dose is the dose determined when the maximum tolerated dose (MTD) cannot be reached.
Time Frame: Within 60 days of Chimeric Antigen Receptor (CAR) T cells infusion
Population: as for outcome 2
Measure: Number; unit: CAR+T cells/kg
Arm/Group | All Participants
Number analyzed (Participants) | 20
CAR+T cells/kg | 0.000006

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 49 months and 19 days.
Description: 6 participants were enrolled but not treated and one participant was enrolled and cells were collected, then came off study because of ineligibility and re-enrolled much later and did receive cells at that time.
Arm/Group | LEVEL 1 - Participants Who Received 0.66x10^6 CAR T Cells Only | LEVEL 1 Foll/by LEVEL 2-Participants Who Received - 0.66x10^6 CAR T Cells Foll/by 2x10^6 CAR T Cells | LEVEL 1 Foll/by LEVEL 3 - Participants Who Received 0.66x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells | LEVEL 2 - Participants Who Received 2x10^6 CAR T Cells Only | LEVEL 2 Followed by LEVEL 3-Participants Who Received 2x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells | LEVEL 3 - Participants Who Received 6x10^6 CAR T Cells Only
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2 | 0/1 | 0/4 | 0/2 | 0/9
Serious Adverse Events (participants affected / at risk) | 3/3 | 1/2 | 1/1 | 3/4 | 1/2 | 8/9
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2 | 1/1 | 4/4 | 2/2 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEVEL 1 - Participants Who Received 0.66x10^6 CAR T Cells Only (N=3) | LEVEL 1 Foll/by LEVEL 2-Participants Who Received - 0.66x10^6 CAR T Cells Foll/by 2x10^6 CAR T Cells (N=2) | LEVEL 1 Foll/by LEVEL 3 - Participants Who Received 0.66x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells (N=1) | LEVEL 2 - Participants Who Received 2x10^6 CAR T Cells Only (N=4) | LEVEL 2 Followed by LEVEL 3-Participants Who Received 2x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells (N=2) | LEVEL 3 - Participants Who Received 6x10^6 CAR T Cells Only (N=9)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (2) | 0 (0) | 2 (4) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — non-invasive follicular thyroid neoplasm with papillary-like nuclear features (nift)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, bacteremia b Fragilis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LEVEL 1 - Participants Who Received 0.66x10^6 CAR T Cells Only (N=3) | LEVEL 1 Foll/by LEVEL 2-Participants Who Received - 0.66x10^6 CAR T Cells Foll/by 2x10^6 CAR T Cells (N=2) | LEVEL 1 Foll/by LEVEL 3 - Participants Who Received 0.66x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells (N=1) | LEVEL 2 - Participants Who Received 2x10^6 CAR T Cells Only (N=4) | LEVEL 2 Followed by LEVEL 3-Participants Who Received 2x10^6 CAR T Cells Foll/by 6x10^6 CAR T Cells (N=2) | LEVEL 3 - Participants Who Received 6x10^6 CAR T Cells Only (N=9)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (3)
Alanine aminotransferase increased (Investigations) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (9) | 2 (7) | 1 (6) | 3 (16) | 2 (7) | 9 (55)
Aspartate aminotransferase increased (Investigations) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (4)
Fever (General disorders) | 3 (8) | 1 (4) | 1 (2) | 3 (6) | 2 (2) | 9 (17)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (10)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2) | 1 (2) | 3 (5) | 1 (1) | 7 (19)
Hyponatremia (Metabolism and nutrition disorders) | 1 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (4) | 2 (7) | 0 (0) | 3 (11) | 2 (4) | 8 (47)
Hypotension (Vascular disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (9) | 2 (17) | 1 (16) | 4 (14) | 2 (13) | 9 (43)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 5 (6)
Neutrophil count decreased (Investigations) | 3 (12) | 2 (10) | 1 (4) | 4 (12) | 2 (15) | 8 (100)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 2 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (13)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 3 (26) | 2 (12) | 1 (9) | 3 (15) | 2 (33) | 9 (101)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck edema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (5) | 1 (2) | 7 (33)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (9)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Mohs surgery (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — squamous cell carcinoma in situ removed from her right shoulder
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 2 (7)
Infections and infestations - Other, Clostridium difficile (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1/1 (2) | 0 (0)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1/1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1/1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/0 (0) | 1 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT02659943/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT02659943/ICF_001.pdf